CLINICAL TRIAL: NCT02667405
Title: The Short Term Effect of Hot Packs and Whirlpool for Increasing Total Active Motion at the Wrist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Mike Szekeres, PhD Candidate, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6712
Record Dates: First submitted 2015-12-07; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures | interventions — Hydrotherapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whirlpool (Experimental): Immersion in Whirlpool during therapy
  Interventions: Procedure: Whirlpool
- Hot Pack (Active Comparator): Hot Pack Application during therapy.
  Interventions: Procedure: Hot Pack

INTERVENTIONS:
Procedure: Hot Pack — Patients have a hot pack and 2 layers of towel wrapped around the wrist and forearm for 15 minutes
  Arms: Hot Pack
Procedure: Whirlpool — Patients immerse their arm, from elbow to hand, in a whirlpool bath of 104 degrees Fahrenheit for 15 minutes
  Arms: Whirlpool

SUMMARY:
This study investigates the effect of hot packs versus whirlpool and exercise for patients with distal radius fracture (DRF). Patients with recently healed DRF are randomized into two groups, with one group receiving hot packs during therapy and the other immersing the arm in a whirlpool for 3 consecutive therapy visits. The effect of these modalities on range of motion and volume of the hand are evaluated, with measurements taking place before and immediately after heat during each visit.

DETAILED DESCRIPTION:
This study investigates the short term effect of hot packs versus whirlpool and exercise for patients with distal radius fracture (DRF) during a therapy visit. Patients with recently healed DRF are randomized into two groups, with one group receiving hot packs during therapy and the other immersing the arm in a whirlpool for 3 consecutive therapy visits.

Measurements of wrist and forearm range of motion, and volume of the hand are recorded before and immediately after heat for each visit, effectively creating six measurement time points. Change scores are recorded for range of motion and for volume, and analyzed using MANOVA to determine differences between groups.

ELIGIBILITY:
Inclusion Criteria:

* Healed DRF,
* allowed to perform motion.

Exclusion Criteria:

* Complex regional pain syndrome,
* inability to read/understand english,
* inability to attend follow up sessions due to driving distance from clinic,
* Raynaud's phenomenon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in Wrist Range of Motion (ROM) | Immediately before and within 5 minutes of completing heat application for 3 consecutive weekly therapy visits
  Measurement of wrist flexion/extension, radial/ulnar deviation/ and pro/supination

SECONDARY OUTCOMES:
Change in Hand Volume | Immediately before, within 5 minutes of completing heat application, then 30 minutes later for 3 consecutive weekly therapy visits
  Volumetric measurement of the hand using a standardized volunteer

CONTACTS AND LOCATIONS:
Overall Officials: Mike Szekeres, PhD (c), Principal Investigator — Western University, Canada
Locations (1):
- Roth McFarlane Hand & Upper Limb Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No